CLINICAL TRIAL: NCT05779306
Title: Performance of Two Sclera Fixated Intraocular Lens Concepts
Acronym: Carlevale
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-011
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cataract Complicated; Cataract Complications Operations
MeSH Terms: conditions — Capsule Opacification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Carlevale: Patients who had a Carlevale lens implanted
  Interventions: Device: IOL Master 700; Device: Casia-2; Device: MS-39; Device: OSIRIS; Device: Autorefractor; Diagnostic Test: Subjective Refraction
- Yamane: Patients who had a lens implanted using Yamane technique
  Interventions: Device: IOL Master 700; Device: Casia-2; Device: MS-39; Device: OSIRIS; Device: Autorefractor; Diagnostic Test: Subjective Refraction

INTERVENTIONS:
Device: IOL Master 700 — Biometry using the IOL Master 700
Device: Casia-2 — Anterior segment-OCT to evaluate lens tilt
Device: MS-39 — Corneal Topography using the MS-39
Device: OSIRIS — Abberometry using the OSIRIS-Abberometer
Device: Autorefractor — Evaluation of Refraction using an Autorefractor
Diagnostic Test: Subjective Refraction — Refraction performed by experienced staff

SUMMARY:
To evaluate and compare the post-operative outcome of two different sceral fixated IOL concepts, the Yamane method (ZA9003, J&J, USA) and the Carlevale IOL (FIL-SSF, Soleko, Italy).

DETAILED DESCRIPTION:
Various approaches to fix the haptics in the sclera can be found in literature. A distinction can be made between suture-fixed and sutureless techniques. The former often proves to be technically challenging and complicated, which has led to an increased rethinking towards sutureless implantation in recent years.

The popular Yamane technique or "flanged IOL fixation" uses a double-needle technique that creates a scleral tunnel and fixates the haptics seamlessly using two 30-gauge needles. However, the haptics must be bent for this purpose Thus, this method is not ideal, since besides from the high degree of manipulation necessary for implantation of the IOL, it is also prone to dislocation and tilt.

A more recent approach is the Carlevale FIL-SSF IOL (Soleko, Italy), which was developed specifically for use in aphakia with a lack of capsular stability. Using two t-shaped anchors, the lens is positioned in two scleral flaps at 180 degrees to each other, without the preparation of a tunnel or excessive manipulation of the haptics. These two self-blocking anchors also provide a great deal of stability. The extent of abberations is also much less with this type of lens implantation, as the fixed position reduces the risk of them. Thus, the Carlevale technique represents a new, potentially superior option for intrascleral fixation.

However, all these types of implantation are not free from aberrations, tilt, or even dislocation. Many factors influence the outcome of IOL implantation, the optimal choice of intraocular lens power, the surgeon's experience regarding fixation in more challenging eyes, or individual anatomical conditions. As part of quality management, an evaluation of monthly and six-monthly data will be performed. The aim of this study is the evaluation of the postoperative tilt of the Carlevale lens, as well as the evaluation of the corrected and uncorrected visual acuity and the anterior chamber depth within the clinical quality management. Patients who have already undergone surgery are called to our clinic by telephone at the earliest 6 weeks after surgery for a one-time follow-up appointment.

The collected data is then evaluated and analyzed as well as compared to the Yamane data.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 21 years
* planned surgery or already taken place surgery using a scleral fixated lens

Exclusion Criteria:

* best corrected visual acuity <0.05 Snellen
* pregnancy
* missing informed consent form

Ages: 21 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients recruited all underwent ocular surgery with implantation of a scleral fixated lens, either using the Carlevale lens or the Yamane technique
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Tilt | 6 Weeks
  Postoperative Tilt
Autorefraction | 6 Weeks
  Refraction using an automated refractor
Subjective Refraction | 6 Weeks
  Refraction performed by experienced staff
Best corrected visual acuity | 6 Weeks
  Measurement performed by experienced staff
uncorrected visual acuity | 6 Weeks
  Measurement performed by experienced staff

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — Johannes Kepler University
Locations (1):
- Department for Ophthalmology and Optometry, Kepler University Hospital GmbH, Johannes Kepler University Linz, Altenberger Strasse 69, 4040 Linz, Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No